CLINICAL TRIAL: NCT04072796
Title: The Effects of Stroke Related Neurogenic Bladder on The Quality of Life: A Study of Turkish Population
Brief Title: Neurogenic Bladder and Quality of Life in Patients With Stroke
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: TURKEYPMR
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Stroke, Complication; Neurogenic Bladder
Keywords: urinary bladder, neurogenic; quality of life; socioeconomic factors; stroke rehabilitation
MeSH Terms: conditions — Stroke; Urinary Bladder, Neurogenic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Case group reported urinary complaints
  Interventions: Behavioral: Questionnaires
- Control group: Control group did not have any urinary complaints.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Short Form-36 (SF-36), Barthel Index (BI), Functional Ambulation Category (FAC), Mini-Mental Test (MMT) and Beck Depression Inventory (BDI) questionnaires

SUMMARY:
This study investigated effects of the neurogenic bladder on the quality of life in stroke survivors. Patients were divided into two groups: the First group consisted of patients with neurogenic bladder and the Second group consisted of patients without neurogenic bladder.

DETAILED DESCRIPTION:
Neurogenic bladder after stroke is a commonly encountered medical condition which slows down the recovery process and exacerbates the functional status of the patient. The neurogenic bladder may possibly affect the quality of life of patients with stroke.

Objectives: The aim of this study is to investigate the relationship between the quality of life and the neurogenic bladder in Turkish stroke survivors.

Methods: 71 patients with stroke were included in the study. Patients were divided into two groups: the First group consisted of patients with neurogenic bladder and the Second group consisted of patients without neurogenic bladder. Short Form-36 (SF-36), Barthel Index (BI), Functional Ambulation Category (FAC), Mini-Mental Test (MMT) and Beck Depression Inventory (BDI) questionnaires were applied to both groups for clinical evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Hemorrhagic or ischemic stroke
* No previous stroke history
* Disease duration > 6 months

Exclusion Criteria:

* Patients with different stroke etiologies other than cerebrovascular events (such as traumatic and tumoral pathologies)
* Previous multiple stroke history
* Pre-stroke urinary complaints
* Previous urogenital surgery history
* Spinal Cord Injury (SCI)
* Prostate volume of > 35ml documented with urinary ultrasonography
* Bladder outlet obstruction
* Poorly controlled Diabetes Mellitus (DM)
* Concomitant neurological diseases such as Multiple Sclerosis and Parkinson's Disease
* Anticholinergic, alpha agonist-antagonist drug use
* Sensory and global aphasia
* Severe communication impairment

Ages: 30 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients who were hospitalised to Istanbul Physical Medicine and Rehabilitation Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Short Form-36 (SF-36) | 15 minutes
  Short Form-36 (SF-36) was used to evaluate the quality of life of the patients. The form consists of 36 items, which measure 8 dimensions. These include (1) Physical function, (2) Social function, (3) Pain, (4) Energy/vitality, (5) Role limitation due to emotional problems , (6) Role limitation due to physical health problems, (7) Mental health and (8) General perception of health. Each subscale is evaluated between 0-100 points. A higher score indicates the better health.

SECONDARY OUTCOMES:
Beck Depression Inventory | 15 minutes
  Beck Depression Inventory was used to assess depressive signs. The scale consists of 21 items and the items are ordered from mild to severe. Evaluation is performed in a range of 0-63 points. The lower score indicates the better psychological profile.
Mini Mental Test (MMT) | 15 minutes
  Mini Mental Test (MMT) was used to evaluate the extent of cognitive impairment. MMT is divided into 5 main categories: orientation (10 points), memory (3 points), attention and calculation (5 points), recalling (3 points) and language (9 points). Total points is 30. Total score between 0-9 points is considered as severe cognitive impairment. Total score between 10-19 points is considered as moderate cognitive impairment. Total score between 20-23 points is considered as mild cognitive impairment. Total score between 24-30 points is considered as normal.
Brunnstrom scale | 15 minute
  Brunnstrom scale is used to evaluate separately upper extremity, lower extremity or hand functions. Six stages are defined. Stage 1: No active movement, Stage 2: Mild spasticity, weak flexor-extensor synergy patterns, Stage 3: Marked spasticity, synergy patterns are evident, Stage 4: Some isolated movements other than synergy patterns can be seen, Stage 5: Decreased spasticity, most muscle activities are isolated, Stage 6: Phasic and well-coordinated isolated movements are performed. A higher point indicates the better status.
Functional Ambulation Category | 15 minute
  Functional Ambulation Category (FAC) was used to evaluate the functional status. FAC assesses human support for ambulation rather than assistive devices. FAC 0: nonfunctional ambulation, FAC 1: Ambulator- dependent for physical assistance level II FAC 2: Ambulator- dependent for physical assistance level I, FAC 3: Ambulator-dependent for supervision FAC 4: Ambulator-independent level surfaces only FAC 5: Ambulator-independent. A higher score indicates the better status.
Barthel Index (BI) | 15 minute
  Barthel Index (BI) evaluates functional independence in term of daily living activity. Total score is 100 points. A higher point indicates better functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye Önes, Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milsom I, Kaplan SA, Coyne KS, Sexton CC, Kopp ZS. Effect of bothersome overactive bladder symptoms on health-related quality of life, anxiety, depression, and treatment seeking in the United States: results from EpiLUTS. Urology. 2012 Jul;80(1):90-6. doi: 10.1016/j.urology.2012.04.004. PMID 22748867
- [Background] Panfili Z, Metcalf M, Griebling TL. Contemporary Evaluation and Treatment of Poststroke Lower Urinary Tract Dysfunction. Urol Clin North Am. 2017 Aug;44(3):403-414. doi: 10.1016/j.ucl.2017.04.007. PMID 28716321
- [Background] Kim KJ, Heo M, Chun IA, Jun HJ; PhDc; Lee JS, Jegal H, Yang YS. The relationship between stroke and quality of life in Korean adults: based on the 2010 Korean community health survey. J Phys Ther Sci. 2015 Jan;27(1):309-12. doi: 10.1589/jpts.27.309. Epub 2015 Jan 9. PMID 25642097
- [Background] Best KL, Ethans K, Craven BC, Noreau L, Hitzig SL. Identifying and classifying quality of life tools for neurogenic bladder function after spinal cord injury: A systematic review. J Spinal Cord Med. 2017 Sep;40(5):505-529. doi: 10.1080/10790268.2016.1226700. Epub 2016 Oct 13. PMID 27734771